CLINICAL TRIAL: NCT01401270
Title: Prize Contingency Management for Cocaine-Dependent Methadone Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sheila Alessi, Associate Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-256-2; R01DA013444 (NIH)
Record Dates: First submitted 2011-07-22; First posted 2011-07-25 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Cocaine Abuse
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment Group A (No Intervention): Standard Care
- Treatment Group B (Experimental): 100% probability of winning a prize with each draw and has 3 prize categories
  Interventions: Behavioral: prize contingency management
- Treatment Group C (Experimental): 31% probability of winning and has 3 prize categories
  Interventions: Behavioral: prize contingency management
- Treatment Group D (Experimental): 100% probability of winning and has 7 prize categories
  Interventions: Behavioral: prize contingency management
- Treatment Group E (Experimental): 31% probability of winning and has 7 prize categories
  Interventions: Behavioral: prize contingency management
- Treatment Group F (Experimental): usual prize contingency management with a 50% probability of winning from 3 prize categories
  Interventions: Behavioral: prize contingency management

INTERVENTIONS:
Behavioral: prize contingency management — Participants earn the chance to win prizes for the targeted behavior, cocaine abstinence.
  Arms: Treatment Group B; Treatment Group C; Treatment Group D; Treatment Group E; Treatment Group F

SUMMARY:
The investigators will randomize 300 cocaine-dependent methadone patients to 1 of 6 conditions: (a) a control group, (b) a contingency management condition that arranges a 100% probability of winning a prize with each draw and has 3 prize categories, (c) a contingency management condition that arranges a 31% probability of winning and has 3 prize categories, (d) a contingency management condition that arranges a 100% probability of winning and has 7 prize categories, (e) a contingency management condition that arranges a 31% probability of winning and has 7 prize categories, or (f) usual prize contingency management with a 50% probability of winning from 3 prize categories. Magnitudes of reinforcement will be identical across conditions, but lower overall probability conditions arrange for greater chances of winning larger magnitude prizes. The investigators expect that the new contingency management conditions will reduce cocaine use relative to the control condition, that 31% probability conditions will decrease drug use relative to 100% conditions, and that 7-prize category conditions will reduce drug use compared to 3-prize category conditions. In addition, the 31%/7-category condition is expected to be most efficacious. Results will be instrumental for further developing prize contingency management to improve outcomes of cocaine-dependent methadone patients.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* current DSM-IV diagnosis of cocaine dependence
* enrolled at the clinic for >3 months
* on a stable dose of methadone (no changes) for >1 month and not requesting a dose alteration
* submitted >1 clinic cocaine positive sample in the last 6 months
* English speaking
* pass a quiz related to understanding the informed consent form

Exclusion Criteria:

* serious, uncontrolled psychiatric illness
* significant cognitive impairment
* in recovery from pathological gambling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
longest continuous period of cocaine abstinence | three months

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M Alessi, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States